CLINICAL TRIAL: NCT05127993
Title: Comprehensive Evaluation of the Passive Talaris Demonstrator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Kevin De Pauw, Prof. Dr., Vrije Universiteit Brussel
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BUN143201526629
Record Dates: First submitted 2021-10-04; First posted 2021-11-19 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Lower Limb Amputation Below Knee (Injury)
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novel prosthesis (Experimental): A unilateral transtibial amputee will conduct experiments with the novel prosthesis followed by experiments with the current prosthesis.
  Interventions: Device: Passive Talaris Demonstrator
- Current prosthesis (Active Comparator): A unilateral transtibial amputee will conduct experiments with the current prosthesis followed by experiments with the novel prosthesis.
  Interventions: Device: Passive Talaris Demonstrator

INTERVENTIONS:
Device: Passive Talaris Demonstrator — The amputee will walk with the passive Talaris Demonstrator, a novel prosthetic foot, designed and built by "Axiles Bionics".

SUMMARY:
The passive Talaris Demonstrator (TD) is developed in continuation of previous prototypes. The main goal of the experiment is to evaluate the effectiveness of TD during daily activities.

DETAILED DESCRIPTION:
Twenty-eight healthy active participants with an unilateral transtibial amputation will conduct 2 experimental trials (EXP1 & EXP2) on the same day in a randomized order, i.e. EXP1 with the currently used prosthesis and EXP2 with the passive Talaris Demonstrator. Each experimental trial will include 6 minutes of treadmill walking at 3 different speeds in consecutive blocks of 2 minutes, a slope walking test, a stair climbing test, a L-test and an outdoor walking task.

The six minutes walk test (6MWT) has become one of the most widely used performance-based outcome measures of functional mobility and exercise capacity. Recently, the 6MWT has been found to correlate with single-limb balance time and symmetry of step length in people with amputation. Additionally, the 6MWT distance has been shown to be responsive to functional training interventions in people with lower-limb amputation. Six minutes of treadmill walking at 3 different speeds will be performed. This test will be performed in consecutive blocks of 2 minutes. These consecutive blocks will be walking 2 minutes at self-selected (SS) speed, 2 minutes at 75% of the SS speed and 2 minutes at 125% of the SS speed. These different walking speeds elicit different angular positions of the ankle and activation levels of muscles, and thus might alter the effectiveness of the novel device.

The slope walking test assesses the participants' ability to ascend and descend a 6 m long ramp of 10% inclination as fast as possible. For safety reasons bilateral handrails are warranted. Participants start the test in an upright position in front of the ramp and are asked to ascend the ramp, turn around on the platform, descend the ramp and return to the starting position.

The stair climbing test assesses the participants' ability to ascend and descend a staircase (84 cm total height, 3-step staircase with an average rise of 28 cm and run of 18 cm). Participants start in front of the staircase and are asked to ascend and descend as fast as possible. Again, bilateral handrails are required to allow support when needed. The ascending phase is initiated with the prosthetic side, while the first step of the descending phase is performed with the non-involved leg.

The L-test, requires higher physical activity of the user. During the L-test, participants are asked to rise from a chair, walk 7 meters, turn 90 degrees, walk 3 meters, turn 180 degrees and then return in the same way to the seated position. A total distance of 20 meter is covered.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transtibial (below knee) amputation
* Unilateral transfemoral (above knee) amputation
* Healthy subject
* Medicare Functional Classification Level: K2-4

Exclusion Criteria:

* Any neurological disease
* Upper limb or bilateral amputation
* Stump pain or bad fit of the socket

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
Performance | Through study completion, a period of 4 months
  Heart rate during all tasks
Performance | Through study completion, a period of 4 months
  Time needed to perform the L-test
Performance | Through study completion, a period of 4 months
  Speed during 6 minutes walk test
Physiological | Through study completion, a period of 4 months
  Electromyography: lower limb muscle activity during different movements (% of the MVC)
Physiological | Through study completion, a period of 4 months
  Oxygen consumption during stair climbing, slope walking and during the 6 minutes walk test
Psychological | Through study completion, a period of 4 months
  Visual analogue scale for comfort (score: 0= not comfortable, 100 = comfortable) and fatigue (score: 0= not fatiguing, 100 = fatiguing) during all tasks
Biomechanical | Through study completion, a period of 4 months
  Joint angels and joint angular velocities of hip, knee and ankle joints

CONTACTS AND LOCATIONS:
Overall Officials: Kevin De Pauw, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Vrije Universiteit Brussel, Brussels, Belgium